CLINICAL TRIAL: NCT05522036
Title: Clinical Evaluation of a Short Illumination Duration (35 Minutes) When Performing Photodynamic Therapy of Actinic Keratosis Using the Dermaris ®
Brief Title: Clinical Evaluation of a Short Illumination Duration (35 Minutes) When Performing PDT of AK Using the Dermaris ®
Acronym: Dermaris-35
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Dermatologique du Roy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR-2022-01
Record Dates: First submitted 2022-07-07; First posted 2022-08-30 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Actinic Keratoses
Keywords: Photodynamic Therapy; Actinic Keratoses; White Light; Methyl ALA
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients treated with Methy ALA & 35 minutes white light illumination (Experimental): Only patients with a minimum of 9 clinically diagnosed grade I and II AK lesions of the scalp (according to the classification by Olsen et al. suggesting the existence of field cancerization, are included in the study. All patients are informed about the purpose of the study and gave informed consent before inclusion. The illumination begins 10 min after the application of MAL cream to the treatment area. In this study, the duration of the light exposure is reduced to 35 min to achieve a PpIX-weighted daylight of 4 J/cm2. MAL cream is removed after the illumination procedure leading to an incubation time of 45 min.
  Interventions: Combination Product: Metvix + Dermaris

INTERVENTIONS:
Combination Product: Metvix + Dermaris — Photodynamic Therapy

SUMMARY:
This clinical study aims aims to evaluate the clinical outcomes of SDL-PDT (simulated daylight Photodynamic Therapy) using the Dermaris in patients treated for AK lesions of the scalp at our medical dermatology center using only 35 minutes low-intensity light exposure.

DETAILED DESCRIPTION:
25 patients, with phototype 1 to 3, with grade I-II AK of the scalp will be treated. Only patients with a minimum of 9 clinically diagnosed grade I and II AK lesions of the scalp (according to the classification of Olsen) suggesting the existence of field cancerization, will treated with SDL-PDT (simulated daylight Photodynamic Therapy) using the Dermaris® (Surgiris, France) and therefore included in the study after application of MAL cream (Metvix ®, Galderma, Switzerland) to the treatment area. After debridment of all treated areas with sandpaper, Metvix will be applied and illuminated with with Dermaris 10 minutes later (leading to drug-light interval (DLI) of 10 minutes) with an irradiance of 2.9 mW/cm2 and a duration of 35 minutes The primary endpoint will be the rate of patients with less than two AK lesions at six-month post-treatment. Secondary endpoints will include scores of pain, erythema, crusts, discomfort and during or/and post the treatment.

A ﬁrst follow-up visit will be scheduled seven days after the treatment. At this visit, crusts will be clinically rated by a dermatologist, while patients scored discomfort they had experienced during the six-day post-treatment. At the second follow-up visit conducted three months after the treatment, AK lesions will be counted by a dermatologist without differentiation between new and recurrent lesions. A second SDL-PDT using the Dermaris will be performed on the day if AK lesions are still present. At last, in case of remaining AK observed at 6 month follow up, a third treatment session with the same parameters will be carried out.

The study is approved by the Ethical clinical committee of the Centre Dermatologique du Roy and conducted in accordance with the ethical principles of the Declaration of Helsinki (2008) and the International Conference on Harmonisation - Good Clinical Practices and in compliance with local regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* phototype 1 to 3,
* grade I-II AK of the scalp
* minimum of 9 clinically diagnosed grade I and II AK lesions of the scalp (according to the classification of Olsen) suggesting the existence of field cancerization

Exclusion Criteria:

* serious organic disorder,
* incipient or established cognitive impairment
* pregnancy
* lactation,
* to be receiving oral or parenteral pharmacological therapy which might interfere with the results.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Lesion clearance rate | 1 year
  The number of removed lesions at six-month post treatment will be expressed as percentage: number of removed lesions divided by number of lesions at patients' inclusion.

SECONDARY OUTCOMES:
Pain & discomfort. | immediately and 6 days after the procedure
  A Visual Analogue Scale (VAS) will be used to measure pain intensity. The VAS consists of a 10cm ruler used to measure the distance in centimeters from the 'no pain marker' (or zero) to the current pain mark. This will provide a pain intensity score out of 10; for example, 6 out of 10 (or 6/10).
  Discomfort during the treatment, which arises from the need for patients to stay under the Dermaris during the 35 minutes of photoactivation, includes joint pain, fatigue, refraining from going to the toilet will be assessed thanks to a specific questionnaire Similarly, discomfort during the six-day post-treatment, which refers to patients' quality of life, includes difficulty to sleep well, inconvenience in head care, embarrassment for outings will be assessed thanks to a specific questionnaire.
Crust & erythema | At 6 days after the procedure
  At six-day post-treatment, the crusts will be rated using a 6-point scale (0 stands for no crusts, 1 for very mild crusts, 2 for mild crusts, 3 for moderate crusts, 4 for severe crusts and 5 for very severe crusts). The presence of an erythema will be noted. 0: no erythema; 1: erythema.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Dermatologique du Roy, Lasne, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be available thanks to an article published in a peer-reviewed open access journal.
Supporting Information: Study Protocol
Time Frame: Individual Participant Data (IPD) will be available 6 months after the completion of the clinical study
Access Criteria: open access journal thanks to a link
URL: https://www.mdpi.com/1424-8247/16/10/1454

REFERENCES:
- [Result] Creusot M, Mordon S. Clinical evaluation of a short illumination duration (1 hour) when performing photodynamic therapy of actinic keratosis using the Dermaris light source. Photodiagnosis Photodyn Ther. 2021 Dec;36:102618. doi: 10.1016/j.pdpdt.2021.102618. Epub 2021 Nov 4. PMID 34743007
- See also: Clinical site — https://www.centredermatologiqueduroy.be/